CLINICAL TRIAL: NCT06889519
Title: A Mentalization-based Intervention to Enhance the Quality of Caregiver-child Interaction and Reduce the Risk of Child Maltreatment: a Pilot Randomized Controlled Trial
Brief Title: Lighthouse Parenting Nanai: a Mentalization-based Group Therapy for Caregivers with History of Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Diego Portales (Other)
Responsible Party: Principal Investigator, Stefanella Costa Cordella, Professor, University Diego Portales
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Fondecyt3220844; 3220844 (Other Grant/Funding Number: ANID (National Agency for Research and Development of Chile))
Record Dates: First submitted 2024-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Child Maltreatment; Trauma, Psychological
Keywords: mentalization-based treatments; , cultural adaptation; child maltreatment; caregiving relationship
MeSH Terms: conditions — Psychological Trauma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, both the participants and the outcomes assessors are blinded to the treatment assignments. Participants are unaware of which one of the interventions are receiving. The outcomes assessors, who are responsible for evaluating the results of the intervention, do not have access to information about which intervention each participant received, ensuring that their assessments are unbiased.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychoeducation Group (Active Comparator): This group receives weekly psychoeducational information
  Interventions: Behavioral: Psychoeducational cards
- MBT Lighthouse NANAI (Experimental): This group receives the psychosocial intervention MBT Lighthouse NANAI
  Interventions: Behavioral: MBT Lighthouse Parenting Program

INTERVENTIONS:
Behavioral: MBT Lighthouse Parenting Program — Lighthouse Parenting Programme, a 12-week intervention for parents, focusing on enhancing mentalizing abilities. It includes weekly group sessions (2hrs) led by 3 trained MBT psychotherapists for 8-12 parents, and fortnightly individual parenting sessions (1hr) with a practitioner. The programme, rooted in Mentalization-Based Treatment (MBT) skills, explores parents mentalizing and their childrens mentalizing and attachment styles through a variety of interactive methods, including multimedia resources and creative activities to stimulate mentalizing. Central to the programme is the metaphor of the parent as a lighthouse, guiding their child. Training for practitioners spanned 4 days, covering MBT and Lighthouse Parenting skills, with an emphasis on experiential learning and self-reflection. Ongoing weekly group supervision will ensure the quality and fidelity of the intervention. Delivered in person at University Diego Portales.
  Arms: MBT Lighthouse NANAI
Behavioral: Psychoeducational cards — They will receive weekly information on parenting in the first 3 years of life. They will have direct contact (via WhatsApp) with a child psychologist to ask questions about the material and to refer to specialized support if needed.
  Arms: Psychoeducation Group

SUMMARY:
The goal of this feasibility randomized controlled trial is to evaluate the effectiveness and acceptability of the Lighthouse Mentalization-Based Treatment Parenting Program (Lighthouse MBT-P) as an intervention for parents at risk of maltreating their children. The study focuses on parents with a history of childhood trauma, aiming to improve parent-child relationships, reduce parenting stress, and ultimately decrease the risk of child maltreatment.

The goal of this study is to test how well the Lighthouse Mentalization-Based Treatment Parenting Program (Lighthouse MBT-P) works for parents who may be at risk of harming their children. The program aims to help parents understand and manage their own and their children's emotions better. By improving these skills, the program hopes to reduce stress in parenting and lower the chances of child abuse or neglect.

The main questions this study will answer are:

* Can parents follow and complete the Lighthouse MBT-P program?
* Does the program help lower stress in parenting and improve relationships between parents and their children?

Participants in this study will:

* Attend weekly group sessions for 12 weeks. These sessions will teach them how to better understand and manage emotions.
* Take part in discussions led by trained psychologists.

Researchers will compare the results of parents who take part in the Lighthouse MBT-P program with those who receive standard parenting support to see which approach works better.

DETAILED DESCRIPTION:
This study is a feasibility randomized controlled trial designed to assess the Lighthouse Mentalization-Based Treatment Parenting Program (Lighthouse MBT-P) for parents who are at risk of maltreating their children. The Lighthouse MBT-P program is specifically tailored for parents with a history of trauma and aims to enhance their mentalizing abilities-helping them better understand and reflect on their own and their children's emotions and thoughts. By improving these skills, the program intends to strengthen parent-child relationships, reduce parenting stress, and ultimately decrease the risk of child maltreatment.

Study Design:

The study is being conducted at Diego Portales University in Santiago, Chile, with a total of 60 participants who will be randomly assigned to one of two groups: the intervention group receiving the Lighthouse MBT-P program and a control group receiving standard psychoeducational support. The intervention will consist of weekly 2-hour group sessions over 12 weeks, where participants will engage in psychoeducation and reflective discussions, facilitated by trained psychologists. These sessions aim to provide parents with the tools to improve their emotional regulation, understand their children's needs better, and develop healthier parenting practices.

Study Phases:

Cultural Adaptation: The Lighthouse MBT-P program has been culturally adapted to ensure its relevance and effectiveness within the Chilean context. This phase involved consultations with local experts, community stakeholders, and pilot testing with a small group of parents to refine the intervention content and delivery methods.

Clinician Training: Therapists who will deliver the Lighthouse MBT-P program have completed a comprehensive training program, including a three-day workshop and ongoing bi-weekly supervision by an MBT specialist. This training ensures that the intervention will be delivered consistently and effectively, adhering to the principles of mentalization-based treatment.

Intervention Delivery: The intervention group will participate in the Lighthouse MBT-P sessions, focusing on enhancing parental mentalizing abilities. The content will cover topics such as emotional regulation, understanding children's behaviors, and managing stress in parenting. Sessions will be conducted online, allowing for greater accessibility for participants.

Data Collection: Data will be collected at multiple time points, including baseline, post-intervention, and follow-up, to assess the feasibility and acceptability of the program, as well as preliminary indicators of its effectiveness in reducing parenting stress and improving parent-child relationships.

Analysis and Interpretation: The data collected will be analyzed using both quantitative and qualitative methods to determine the feasibility of the program and to identify any barriers or facilitators to its implementation. The results will inform decisions about whether to proceed with a full-scale randomized controlled trial and guide any necessary adjustments to the program.

Significance:

This study addresses a critical gap in the availability of trauma-informed, attachment-based interventions for parents at risk of child maltreatment in Chile. By evaluating the feasibility of the Lighthouse MBT-P program, this research aims to provide a foundation for larger-scale interventions that could significantly impact the prevention of child maltreatment and improve the well-being of vulnerable families.

ELIGIBILITY:
Inclusion Criteria:

1. Biological parents of children (0-36 months old) with custody of their child.
2. Parents who have gone through adverse childhood experiences, have a history of parental substance abuse or incarceration, have current exposure to relationship violence, or social isolation, or have lost custody of a child in the past.
3. Parents must be over the age of 18.

Exclusion Criteria:

1. Parents who are unable to provide informed consent due to mental or cognitive impairment,
2. Parents not fluent in Spanish.
3. Child's diagnosis of autistic spectrum disorder or severe cognitive delay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-17 (Actual); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Conducting a Full-Scale Trial: Recruitment, Retention, and Protocol Acceptability Assessed Through Semi-Structured Interviews and Attendance Records | Measured continuously from the start of recruitment through the end of the intervention period (12 weeks for control group, 26 weeks for intervention group).
  The feasibility of conducting a future full-scale trial will be assessed through the following measures:
  Participant Acceptability: Assessed via semi-structured interviews to capture participants' understanding, views, and experiences, including potential barriers or facilitators.
  Clinician Acceptability: Evaluated through in-depth interviews with clinicians, focusing on barriers, facilitators, and perceptions of the intervention.
  Adherence: Monitored through attendance records, with successful adherence defined as at least 65% of participants attending 40% or more of sessions.
  Recruitment and Retention: Recruitment tracked by the percentage of invited participants who consent to participate, with retention determined by the attrition rate, targeting no more than 20%.

SECONDARY OUTCOMES:
Change in Parenting Stress from Baseline to 6-Month Follow-Up Using the Parenting Stress Index-Short Form (PSI-SF) | Measured at three specific points: baseline (pre-intervention), end of treatment (12 weeks for control group/26 weeks for intervention group), and 6-month follow-up.
  Parenting stress will be measured using the Parenting Stress Index-Short Form (PSI-SF), a 36-item self-report questionnaire. The PSI-SF includes three subscales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child, with a Total Stress Score. The minimum score is 36, and the maximum score is 180, with higher scores indicating greater stress. The primary analysis will focus on changes from baseline to the 6-month follow-up after randomization.
Change in Quality of Life in Parents from Baseline to 6-Month Follow-Up Using the SF-36 Health Survey | Measured at three specific points: baseline (pre-intervention), end of treatment (12 weeks for control group/26 weeks for intervention group), and 6-month follow-up.
  The quality of life in parents will be assessed using the SF-36 Health Survey, focusing on the Mental Component Summary (MCS) score. The SF-36 includes 36 items across eight domains, with a scoring range from 0 to 100 for each domain, where higher scores represent better health-related quality of life. The primary analysis will track changes in the MCS score from baseline to the 6-month follow-up after randomization.

OTHER OUTCOMES:
Change in Parental Mentalizing from Baseline to 6-Month Follow-Up Using the Parental Development Interview - Reflective Functioning (PDI-RF) | Measured at three specific points: baseline (pre-intervention), end of treatment (12 weeks for control group/26 weeks for intervention group), and 6-month follow-up.
  Parental mentalizing will be assessed using the Parental Development Interview - Reflective Functioning (PDI-RF), a semi-structured interview that evaluates a parent's capacity to reflect on their own and their child's mental states. Scores range from 1 to 9, with higher scores indicating greater reflective functioning. The study will examine changes in PDI-RF scores from baseline to the 6-month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- University Diego Portales, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
data dictionaries available to other researchers after the end of the study
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: July 2024 to July 2029
Access Criteria: a proposal that describes planned analyses must be submitted and a data sharing agreement must be signed, contacting the principal investigator by e-mail.
URL: https://cepps.udp.cl/